CLINICAL TRIAL: NCT06991387
Title: Exploring the Short-Term Effects of Myofascial Release in Text Neck Syndrome
Brief Title: Acute Effects of Myofascial Release in Individuals With Text Neck Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ece ACAR, Director, Karabuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: text neck syndrome
Record Dates: First submitted 2025-05-20; First posted 2025-05-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Text Neck Posture; Neck Pain; Myofascial Release Technique
Keywords: Text Neck Syndrome; Neck Pain; Myofascial Release
MeSH Terms: conditions — Neck Pain | interventions — Myofascial Release Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants with text neck syndrome (Experimental)
  Interventions: Other: Myofascial Release

INTERVENTIONS:
Other: Myofascial Release — A single session of myofascial release techniques including Single Arm Pull, Lateral Neck Shoulder Release, Thoracic Transverse Release, and Anterior Cervical Release applied by a physiotherapist trained in manual therapy.
  Other Names: Manual Therapy

SUMMARY:
This study aims to investigate the acute effects of myofascial release therapy on neck pain, functional status, and cervical range of motion in individuals diagnosed with Text Neck Syndrome (TNS). Text Neck Syndrome is increasingly prevalent due to excessive use of smartphones and other digital devices, particularly among young adults. The intervention will consist of a single session of standardized myofascial release techniques applied to the cervical and thoracic regions. The primary outcome will be neck pain intensity measured using the Numeric Rating Scale (NRS-11), while secondary outcomes will include cervical range of motion and the modified Neck Disability Index (NDI). Assessments will be performed immediately before and after the intervention. The study will be conducted with volunteer participants between the ages of 18 and 40, who use mobile devices for more than 3 hours per day and meet the diagnostic criteria for TNS

DETAILED DESCRIPTION:
Text Neck Syndrome (TNS) is a repetitive stress injury caused by prolonged forward head posture, often due to extended use of mobile phones, tablets, and computers. The increasing prevalence of this postural disorder has led to a rise in musculoskeletal complaints, particularly among young adults and university students. TNS is characterized by symptoms such as neck and upper back pain, stiffness, shoulder pain, headaches, and, in some cases, paresthesia in the upper limbs.

Myofascial release (MFR) is a manual therapy technique aimed at releasing restrictions in the myofascial system to alleviate pain and improve function. It is increasingly being used to treat various musculoskeletal disorders, including those affecting the cervical and thoracic spine. The technique involves applying gentle, sustained pressure to the myofascial connective tissue to improve mobility, reduce pain, and enhance functional performance.

This single-arm experimental study is designed to evaluate the acute effects of a one-time standardized myofascial release session targeting the cervical and upper thoracic regions in individuals diagnosed with Text Neck Syndrome. Four myofascial techniques will be applied in a specific sequence:

Single Arm Pull

Lateral Neck Shoulder Release

Thoracic Transverse Release

Anterior Cervical Release

These techniques are performed by a licensed physiotherapist with advanced training in manual therapy. Each intervention is applied bilaterally (if appropriate), with a duration of 90-120 seconds per technique.

The primary focus is to observe immediate (pre-post) changes in:

Subjective neck pain intensity

Functional disability associated with the neck

Cervical range of motion (C-ROM) in multiple planes

This study is exploratory in nature and aims to provide preliminary data on the efficacy of a single-session MFR intervention for individuals experiencing TNS-related symptoms. The findings may guide future controlled trials and inform physiotherapeutic approaches in addressing posture-related neck dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years (inclusive)
* Uses a mobile device for ≥3 hours/day
* Reports at least 3 out of the following 6 symptoms associated with Text Neck Syndrome (TNS):

Neck pain Shoulder pain Back pain Headache Insomnia Numbness/tingling in hands

-Voluntarily agrees to participate and provides informed consent

Exclusion Criteria:

* History of congenital, traumatic, or surgical pathology affecting the cervical -------spine or shoulder region
* Neurological disorders that cause headaches (e.g., migraines due to underlying neurological conditions)
* Presence of inflammatory, infectious spinal diseases, or diagnosed spinal deformities
* Received trigger point injections in the cervical region within the past 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Baseline and immediately post-treatment
  Change in neck pain intensity using the 11-point NRS (0=no pain, 10=worst possible pain)
Cervical Range of Motion and joint position sense | Baseline and immediately post-treatment
  Measured using a phone application (Clinometer) for flexion, extension, rotation, and lateral flexion

SECONDARY OUTCOMES:
Modified Neck Disability Index | Baseline and immediately post-treatment
  Assessment of disability related to neck pain (score range: 0-50)

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük University, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grasser T, Borges Dario A, Parreira PCS, Correia IMT, Meziat-Filho N. Defining text neck: a scoping review. Eur Spine J. 2023 Oct;32(10):3463-3484. doi: 10.1007/s00586-023-07821-2. Epub 2023 Jul 5. PMID 37405530
- [Background] Mishra D, Prakash RH, Mehta J, Dhaduk A. Comparative Study of Active Release Technique and Myofascial Release Technique in Treatment of Patients with Upper Trapezius Spasm. J Clin Diagn Res
- [Background] Gauns SV, Gurudut PV. A randomized controlled trial to study the effect of gross myofascial release on mechanical neck pain referred to upper limb. Int J Health Sci (Qassim). 2018 Sep-Oct;12(5):51-59. PMID 30202408